CLINICAL TRIAL: NCT04797676
Title: Different Methods of Pancreatic Ductal Adenocarcinoma Specimen Acquisition, EUS-FNB vs. Surgery, Influence on Culturing Primary Cells to Screen Sensitive Chemotherapeutics for Individuals: a Prospective Cohort Study
Brief Title: Effects of Different Methods of PDAC Specimen Acquisition on Primary Cell Culture and Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021EUS-002
Record Dates: First submitted 2021-03-01; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators use two methods (EUS-FNB and surgery) to obtain pancreatic cancer specimens from patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS-FNB group: Each patient participated in the EUS-FNB group and the surgery group. The procedure of EUS-FNB with wet suction technique is as follow: before the needle was inserted into the biopsy channel, the stylet was removed, and the needle was flushed with saline solution until the fluid dripped out of the needle tip. The air column was replaced with the fluid. A 10-mL syringe was prefilled with 2 mL of saline solution, and the valve was closed. The syringe was loaded to the 5-mL position (i.e. a 3-mL vacuum) and then attached to the proximal port and used for biopsy after inserting into the biopsy channel and puncturing the lesion. Each patient was performed 1-2 passes to obtain specimens for subsequent experiments.
  Interventions: Procedure: different methods of specimen acquisition
- surgery group: Each patient participated in the EUS-FNB group and the surgery group. The patient underwent EUS-FNB with wet suction technique first, followed by surgery (palliative surgery without excising tumor is not included) for pancreatic cancer. According to the size of the specimen, 0.5cm3-1cm3 tumor specimen was used for subsequent experiments.
  Interventions: Procedure: different methods of specimen acquisition

INTERVENTIONS:
Procedure: different methods of specimen acquisition — After informed consent, the investigators use two methods to obtain specimens for patients with pancreatic ductal adenocarcinoma, who needs eus-fnb for auxiliary diagnosis and had the opportunity of surgery. One method is EUS-FNB with wet suction technique, the other is surgery (including radical operation and cytoreductive surgery). Both methods are used on the same patient to remove deviations in results caused by tumor heterogeneity.

SUMMARY:
The purpose of this study is to investigate the difference in the success rate of culturing primary cells derived from pancreatic ductal adenocarcinoma specimens of patients which obtained by endoscopic ultrasound-guided fine-needle biopsy wet suction technique and surgery, analyze whether the sensitive chemotherapeutic agents screened by the primary cells cultured from the specimens obtained by the above two methods are consistent, and whether they are consistent with the clinical treatment effect of patients, verify the accuracy of laboratory drug sensitivity results, so as to provide the basis for pancreatic ductal adenocarcinoma patients to choose the source of individual treatment samples.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the malignant tumors with the highest mortality rate in the world, with a 5-year survival rate of only 7.2%-9%. Because some patients are resistant to multiple chemotherapy drugs, and there are differences in drug sensitivity between individuals, the current pancreatic ductal adenocarcinoma (PDAC) chemotherapy effect is not satisfactory. In order to improve the efficacy of chemotherapy and achieve precise treatment, it is important to establish an accurate and individualized PDAC research model.

At present, several studies have reported that surgical specimens of pancreatic cancer are successfully used to cultivate preclinical research models. However, most patients with PDAC have developed to advanced stage at the time of diagnosis and are not suitable for surgery, which limits our ability to obtain tumor cells. Endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) can procure specimens when patients have not receive any treatment, and can also evaluate the therapeutic effect and tumor progression in the process of treatment.

Until now, there is no study to compare the efficiency of the two methods in constructing preclinical research model of pancreatic cancer. Therefore, the investigators intend to investigate the difference in the success rate of culturing primary cells derived from PDAC specimens of patients which obtained by EUS-FNB wet suction technique and surgery, analyze whether the sensitive chemotherapeutic agents screened by the primary cells cultured from the specimens obtained by the above two methods are consistent, and whether they are consistent with the clinical treatment effect of patients, verify the accuracy of laboratory drug sensitivity results, so as to provide the basis for PDAC patients to choose the source of individual treatment samples.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥18
2. Imaging examination (US, MRI, CT or PET-CT) of patients confirmed pancreatic lesions, and considered the possibility of PDAC, EUS-FNB was needed for auxiliary diagnosis
3. No chemotherapy, including neoadjuvant chemotherapy, postoperative adjuvant chemotherapy and palliative chemotherapy, has been performed on patients
4. Having surgery opportunities (including radical operation and cytoreductive surgery) and willingness of operation
5. Agree to attend this study and signed informed consent

Exclusion Criteria:

1. Poor physical condition, including but not limited to hemoglobin ≤ 8.0g/dl, severe cardiopulmonary insufficiency, etc
2. Coagulation dysfunction (platelet count < 50,000/mm3, international standardized ratio > 1.5), or inability to discontinue anticoagulation therapy
3. High risk for deep sedation
4. Acute pancreatitis in the previous 2 weeks
5. Pregnancy or lactation
6. Any diseases leading to unreliable follow-up
7. Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are considered as PDAC by imaging, and may have opportunity of surgery, and require EUS-FNB for definite diagnosis will potentially be included in this study. Informed consent will be given by the doctor in charge or endoscopic operator or researcher. Patients who agree to participate in the trial will sign an informed consent form. Patients were enrolled after being screened according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The different culture success rate | About 6 weeks after operation
  The difference in the success rate of primary cell culture (P1) and passage to the third generation (P3) between PDAC specimens obtained by EUS-FNB and those obtained by surgery.
The representation of the primary cells of pancreatic cancer | About 8 weeks after operation
  Through Western Blot and PCR methods to detect the representativeness of primary cells to the primary tumor. If the patient underwent surgery later, hematoxylin-eosin staining and/or immunohistochemistry were added to compare the histological morphology with the original tumor.

SECONDARY OUTCOMES:
Differences in drug susceptibility results between the two groups | About 14 weeks after operation
  The primary cells cultured from PDAC which obtained by two methods, EUS-FNB and surgery, are used to screen sensitive chemotherapeutic drugs commonly used in pancreatic ductal adenocarcinoma, and to see if there are any differences between the two groups.
Differences of drug sensitivity results between in vitro and clinical drug results | About 22 weeks after operation
  The results of the commonly used sensitive chemotherapeutics for pancreatic ductal adenocarcinoma screened by the two groups of primary cells are fed back to the clinician. If the patients have not started chemotherapy, the drug will be used according to the results screened in vitro to observe whether the tumor markers improved and the tumor size decreased. If the patients have completed chemotherapy, the laboratory results are compared with the clinical results of chemotherapy, i.e., whether the in vitro screening results of sensitive/resistant drugs have the same effect in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, M.D., Principal Investigator — The Third Xiangya Hospital, Central South University
Locations (1):
- The Third Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No